CLINICAL TRIAL: NCT01902095
Title: Evaluation of the Clinical Effects of Tooth Powder on Plaque Induced Gingivitis
Brief Title: Clinical Effects of Tooth Powder on Gingivitis
Acronym: Toothpowder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Collaborators: Fatima Jinnah Dental College (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Khalil Khan, Associate Professor, Sheikh Zayed Federal Postgraduate Medical Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KhanMK-2012
Record Dates: First submitted 2013-05-09; First posted 2013-07-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-05

CONDITIONS: Gingivitis; Mouth Diseases
Keywords: tooth pastes; tooth powders; Stain Index
MeSH Terms: conditions — Gingivitis; Mouth Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tooth powder (test) arm (Experimental): Experimental arm: tooth powder
  Interventions: Device: Tooth powder
- Tooth Paste (control) (Active Comparator): Tooth Paste
  Interventions: Device: Tooth paste (control)

INTERVENTIONS:
Device: Tooth powder — Each participant was handed over a sealed pack containing a teeth cleaning kit that included tooth powder (test) or toothpaste (control) and a new soft toothbrush along with written and verbal instructions of usage. They were advised to brush their teeth twice a day with the given dentifrices and tooth brush for two weeks.
  Arms: Tooth powder (test) arm
Device: Tooth paste (control) — Active Comparator
  Other Names: Tooth paste
  Arms: Tooth Paste (control)

SUMMARY:
Dental plaque, known as dental biofilm, is implicated as the primary etiological agent responsible for oral inflammatory diseases. Matured form of dental plaque plays a major role in the pathogenicity of gingivitis; if not managed in early stages it results in a cascade of events leading to the destruction of periodontal tissues.

Effective plaque control techniques have been suggested that maintain dental biofilm at levels compatible with oral health and is the cornerstone for all preventive strategies to control oral diseases particularly gingivitis. To clean teeth and ensure effective plaque control, different mechanical means have been in use since centuries. However because of an inadequacy in plaque removal, different antimicrobial and antiplaque agents have been introduced in oral-care products.

The use of dentifrices has been recommended over the years as the ultimate way of preventing the incidence of oral diseases. Dentifrices have the anti-plaque and the anti-gingivitis capabilities due to their composition. Toothpastes and to a lesser extent toothpowders are common oral-care products used to eliminate plaque and other deposits from tooth surfaces. Existent literature has focused more on toothpaste and mouth rinse and derelicts toothpowder despite its difference owing to the absence of humectants. With the intention to advance the knowledge on this issue as well as close the research gap, this study was conducted to evaluate the efficacy of toothpowder in alleviating gingivitis, controlling dental plaque, and inhibiting extrinsic stains.

A single-blind, parallel arm randomized controlled trial (RCT) evaluated the efficacy of toothpowder against toothpaste through oral hygiene parameters of plaque and stain deposits on teeth and gingival inflammation. Plaque Index, Lobene Stain Index and Gingival Index were used as measures of oral hygiene.

The current RCT revealed that toothpowder and toothpaste were equally effective in both treatment and control groups from clinical perspective however toothpowder showed a statistically significant effectiveness as compared to toothpaste. Toothpowder, composed of calcium carbonate and essential oils, has demonstrated to be statistically more effective than toothpaste in controlling extrinsic dental staining, dental plaque and gingival inflammation.

DETAILED DESCRIPTION:
A single-blind randomized controlled trial was conducted during November 2010 and October 2011. After screening and consent, eligible subjects received mechanical periodontal therapy. Subjects were then randomized to Test group and Control group at a 1:1 ratio. The test group was provided tooth powder and a control group received toothpaste. Healthy subjects with plaque induced gingivitis and who fulfilled the inclusion criteria were recruited from the Department of Periodontology, Fatima Jinnah Dental College Hospital, Karachi, Pakistan.77 subjects with gingivitis were randomized to test group and 77 subjects to the control group. Therefore, to complete the randomized controlled trial, a total of 154 subjects were recruited and randomized.

Outcome measure gingivitis was measured through plaque index, gingival index and Lobene stain index.

ELIGIBILITY:
1. Inclusion Criteria

   1. Male or female
   2. Age ≥ 18-to-65 years (18th birthday completed)
   3. In good general health
   4. Available for the duration of the study
   5. Able and willing to follow study protocol
   6. Able and willing to sign approved informed consent
   7. At least 20 natural teeth suitable for evaluation
   8. Full mouth Gingival Index (GI) score ≥ 1.04
2. Exclusion Criteria

   1. Females disagree to birth control measure for the duration of the study
   2. Having any acute /chronic systemic illness
   3. Current smokers or tobacco users
   4. Pregnant or lactating Females
   5. Allergy to the ingredients of the products to be tested
   6. Requiring pre-medication prior to dental appointment
   7. Antibiotic use in the last 3 months
   8. Routine use of anticoagulant medication
   9. Routine use of anti-inflammatory medication
   10. Routine use of medications known to have effects on the gingiva e.g., phenytoin etc)
   11. Routine use of medications inhibiting or stimulating salivary flow
   12. Physical handicap that could interfere with daily performance of oral hygiene
   13. Participation in any other study during the study period of this trial
   14. Routine use of any mouthrinse
   15. Routine use of any interdental cleaning device (floss, dental toothpicks)
   16. Having any removable appliance
   17. Having fixed orthodontic appliances (including permanent orthodontic retainers)
   18. Having probing depth ≥4 mm at any site
   19. Having had active periodontal therapy during the last 6 months
   20. Had periodontal prophylaxis or periodontal maintenance therapy in the last 3 months
   21. More than 3 carious lesions requiring immediate care
   22. Gross oral pathology (e.g., tumors, candidiasis, mucocutaneous disease)

Ages: 33 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Gingivitis | November 2010 - October 2011 (up to 1 year)
  Gingival Index (Löe and Silness, 1963) modified by Talbott et al. (1977) was used for the assessment of the gingival condition and record qualitative changes in the gingiva. Its scores (0 to 3) recorded the marginal and interproximal tissues separately. The criteria are: 0= normal gingiva, 1= mild inflammation - slight change in color and slight edema but no bleeding on probing, 2= moderate inflammation - redness, edema and glazing, bleeding on probing and 3= severe inflammation - marked redness and edema, ulceration with a tendency to spontaneous bleeding.

SECONDARY OUTCOMES:
Plaque | November 2010 - October 2011 (up to 1 year)
  Quigley-Hein (Tuersky) Index was used for plaque deposits. This index is based on the visually check of non-restored surface of all the teeth except third molars; this is done on a scale from score 0 to score 5. An index for the entire mouth is determined by dividing the total score by the number surfaces examined. The criteria for scoring are: 0 = no plaque, 1 = separate flecks of plaque, 2 = continuous band of 1 mm, 3 = >1mm and <1/3 of tooth surface, 4 = >1/3 and <2/3 and 5 = >2/3 of tooth covered with plaque
External tooth stains | November 2010 - October 2011 (up to 1 year)
  Lobene index based on the intensity and area of stains covered on the labial surfaces of the anterior teeth was used. Buccal surfaces of teeth are divided into two gingival crescent and body. In this index intensity and area measured on gingival crescent and body separately and also in combination by multiplying intensity and area. An index for the entire mouth is determined by dividing the total score by the number surfaces examined

CONTACTS AND LOCATIONS:
Overall Officials: Ayyaz A Khan, PhD, Study Director — University of the Punjab